CLINICAL TRIAL: NCT02051894
Title: NeoAdapt 3: An Observational Study Investigating Novel Biomarkers in the Evaluation and Treatment of Neonatal Circulatory Insufficiency in Infants Suffering From Hypoxic Ischemic Encephalopathy.
Brief Title: NeoAdapt 3: Novel Biomarkers in the Evaluation of Neonatal Circulatory Insufficiency in Babies Suffering From Hypoxic Ischemic Encephalopathy
Status: Completed | Type: Observational
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Dr Liam Mahoney, Clinical Research Fellow in Paediatrics, Brighton and Sussex University Hospitals NHS Trust
Other Study IDs: IRAS: 145271
Record Dates: First submitted 2014-01-27; First posted 2014-01-31 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Circulatory Failure
Keywords: Neonates; Dobutamine; Superior Vena Cana Flow; Hypoxic Ischemic Encephalopathy; Pleth Variability Index
MeSH Terms: conditions — Shock; Hypoxia-Ischemia, Brain | interventions — Dobutamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Two blood samples of 400µl each will be obtained for each infant receiving dobutamine.
  Samples for the pharmacokinetic studies will utilise micro assays to minimise the amount of blood taken and will coincide with the taking of clinically indicated sample to reduce the burden placed on neonates included in this study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIE Group
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Dobutamine — Infants will receive treatment according to the preference of the responsible physician. As is common practice, dobutamine, dopamine and/or other treatments (including other cardiovascular drugs and/or volume replacement therapy with normal saline) will be administered.
  If dobutamine is used we will take a maximum of two blood samples from the baby for pharmacokinetic analysis.

SUMMARY:
1 in 1000 babies are born suffering from a lack of oxygen. This is known as hypoxic ischemic encephalopathy (HIE). Infants with this condition can suffer multiple organ problems. In particular it can affect how their hearts pump blood around their body thus leading to a poor blood supply to parts of their body such as the brain. This is known as circulatory failure and can contribute to poor long term outcomes such as cerebral palsy. To try and prevent brain damage these infants are treated with total body cooling, however this treatment can further effect how babies pump blood around the body, but also how drugs which may be used by in this condition are processed.

In order to assess and treat this condition doctors need to be able to accurately measure the blood supply in an infant. However there is no agreement on how best to do this. This makes decisions about when to treat an infant difficult. Sometimes doctors may want to use drugs such as dobutamine or adrenaline but these drugs are unlicensed in babies.

This study proposes to observe the way babies circulatory problems are treated in babies with HIE the in the first four days of life. In addition the study will look are two new measurements of a babies blood supply to see if they are a better measure of when an infant needs treatment. This will involve an ultrasound scan of the heart and measurement of the baby's oxygen levels from a probe placed on their hand. The study will also look at how the drug dobutamine is processed by babies. This will be done from two small extra blood tests. The aim of the study is to help clinicians refine the identification and treatment of circulatory failure in babies with HIE.

DETAILED DESCRIPTION:
The current definitions of neonatal shock/circulatory failure are outdated, inaccurate and it is not be appropriate to apply to infants suffering from hypoxic ischemic encephalopathy he purpose of the this research is to look at older than 33 weeks gestational age in order to fill the knowledge gap here and help in the development a new definition of neonatal circulatory failure.

The main research questions are:-

1. To investigate new non-invasive methods of assessing an infants circulatory status in infants suffering from HIE.
2. To gain initial data on how dobutamine is processed by babies when they are used for circulatory failure.
3. To observe how physicians decide to treat circulatory failure in infants suffering from HIE.

Research has shown that there is up to a 14 fold difference in how doctors assess and treat circulatory failure. In infants suffering from hypoxic ischemic encephalopathy this is complicated further by the fact that treatment with total body cooling can interfere further with how the body pumps blood around the body. This is further complicated by the fact there is no agreed definition for circulatory failure in infants. By investigating new methods of assessing a babies circulatory status we intend to help create a new definition of circulatory failure which will in turn help doctors create further studies to identify infants with circulatory failure and find the best ways of treating this condition in babies. So far research in this area has been concentrated in babies born at less than 33 weeks gestation. We extend the knowledge in the area to infants older that 36 weeks gestation suffering from hypoxic ischemic encephalopathy.

Dobutamine is a drug that does not have a license for use in infants. In the future all new drugs will need to be studied in children before a license for them is given. In addition the European Community are encouraging that research is undertaken to look into the use of old drugs in which are used in babies. As mentioned previously there is very little data to show how dobutamine is handled by babies and contribute to new information on how this drug should be given safely.

This will be an observational pilot study, to gain novel values of SVC flows and pleth values in infants with HIE being treated with total body cooling. In addition this population will be observed with regard to which diagnostic measures that lead to treatment decisions, especially with regards to haemodynamic stability, and what the effect of those decisions are on the various diagnostic measures. Decision-making for their treatment will be based on clinical guidelines in at the Trevor Mann Baby Unit and clinician preference.

The assessment of SVC flow and PVI will only be done every 24 hours whist the infant is receiving total body cooling and once during the re-warming phase of their treatment.

Primary Outcome Measure Values for SVCF and PVI in neonates with HIE admitted for total body cooling derived from Echo-D and plethysmographic studies .

Observed Clinical Outcome Measures

* MRI appearances
* Cranial US appearances
* CFM appearances The MRI will be reported and scored according to a system described by Rutherford et al to aid predict long term outcome. This will be performed within the first two weeks post-total body cooling treatment which is in keeping with national and local guidance.

The analysis of the findings on cranial ultrasound scan will be interpreted in the light of a baseline scan, to be performed as soon as possible after birth on enrolment, to avoid ascribing the effect of antenatal insults to postnatal events.

Those treated for HIE with total body cooling will have an additional daily neurological assessment during the cooling and re-warming phases of treatment that will be a graded according to criteria set out by Sarnat et al. This is routine in the treatment of this population of infants.

CFM recordings will be made during the cooling treatment phase of an infant. This is a standard observation in children with HIE and is associated with long term outcomes for these infants. For the purposes of the study the CFM will be used at the discretion of the attending medical team. The analysis of the CFM will follow what was used in the Toby Trial and is described in detail elsewhere.

Treatments for Circulatory Failure Infants will receive treatment according to the preference of the responsible physician. As is common practice, dobutamine, dopamine and/or other treatments (including other cardiovascular drugs and/or volume replacement therapy with normal saline) will be administered.

Dose of administration The dose of administration of dobutamine will be at the discretion of the responsible physician. We envisage that dobutamine will typically be started between 2.5 and 5 mcg/kg/min and increased in steps of 5 mcg/kg/min to a maximum of 20 mcg/kg/min with a given time frequency if no response is seen.

Any changes to the treatment strategy will be documented by the responsible physician.

Criteria for Up-Titration of Medication Dose escalation will be guided by clinical judgment. Clinicians will be asked to record the criteria they used in order to make this decision.

Criteria for Down-Titration Dose reduction will be guided by clinical judgment. Clinicians will be asked to record the criteria they used in order to make this decision.

Further treatment If there is no response to dobutamine at 20 mcgg/k/min or the clinical response is considered by the attending physician to be inadequate, further treatment will be at the discretion of the attending physician who will be asked to record the reasons for the change in treatment strategy as well as the additional treatment that is given to the patient.

Concomitant therapy There will be no per-protocol concomitant medication or treatment. Accordingly, other important co-interventions will follow specific centre protocols and will be recorded in the case record form.

PHARMACOKINETICS (PK) SUB-STUDY

Aim of the PK sub-studies The aim of the sub-study is to give preliminary information in order to try and construct a population PK model. Given the uncertainties regarding the PK of dobutamine in infants receiving total body cooling we shall assess its elimination half life. This is defined as the amount of time for the quantity of a concentration to fall by half.

Half-life sub-study We will perform a preliminary study on all the infants included in NeoAdapt 3 that receive dobutamine as treatment for haemodynamic insufficiency. Two blood samples, of 400 μl each, will be obtained from each of these patients. The first sample will be drawn after the end of the infusion, at the time when dobutamine ceases reaching the systemic circulation of the neonate, defined as time end (te).

The second sample will be taken at different study time points after the end of infusion:

* 5 min after te
* 15 min after te
* 45 min after te
* 2 hours after te
* 6 hours after te Two infants will be allocated to each time point. Sampling times will be assigned randomly to the patients.

Plasma samples will be sent to the laboratory for the quantification of dobutamine.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the NICU with HIE for total body cooling therapy
* Postnatal age <72 hours
* Parental informed consent

Exclusion Criteria:

* Non-viability
* Congenital hydrops or malformations likely to affect cardiovascular adaptation
* Surgery planned within 72 hours of birth
* Chromosomal anomalies
* Informed consent form (ICF) not signed

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants older than 36 weeks gestational age suffering from hypoxic ischemic encephalopathy receiving total body cooling
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Superior Vena Cava Flow (SVCF) in babys recieving total body cooling for Hypoxic Ischemic Encephalopathy | Once a day for a maximum of three days after birth
  After consent and enrolment, Echo-D assessments will be repeated every 24 of cooling treatment (first 72 hours of postnatal life) and once during the re-warming phase (typically taking 8 hours after cooling has finished). The change in this measurement over the cooling treatment will be recorded.
Pleth Variability Index (PVI) in infants undergoing total body cooling treatment for hypoxic ischemic encephalopathy | Once a day for a maximum of three days after birth
  After consent and enrolment PVI assessments will be repeated every 24 of cooling treatment (first 72 hours of postnatal life) and once during the re-warming phase (typically taking 8 hours after cooling has finished). The changes in the PVI measurements will be recorded over the course of cooling therapy.
Pharmacokinetic data for the emilmination half life of dobutamine when this drug is given for circulatory failure | If dobutamine is given to an infant in the first three days of life
  If dobutamine is given for circulatory insufficiency in the first three days of life 2 blood samples will be taken for pharmacokinetic analysis of dobutamine.

SECONDARY OUTCOMES:
SVCF and PVI values corrleation to each other and to parameters that assess circulatory status such as mean blood pressure and capillary refill time | Over the first 3 days of life
  Correlation analysis will be used to determine if there is an association between SVCF and PVI values to common parameters that are used in the neonatal intensive care setting to assess the haemodynamic status of an infant.
SVCF and PVI values relationship to clinical outcomes | Over the first three days of life
  Clinical outcomes for infants who are suffering from hypoxic ischemic encephalopathy, such as MRI appearances, will be recorded. These outcomes will be compared to the SVCF and PVI values gained to see if either measurement is predictive of such clinical outcomes.
SVCF and PVI values and dobutamine treatment for circulatory failure | Over the first three days of life
  Comparisons between the will be made between SVCF and PVI values gained from infants who were and those who were not receiving dobutamine at the time of these measurements to see if there is a significant difference between the values gained.

CONTACTS AND LOCATIONS:
Overall Officials: Liam Mahoney, B, Principal Investigator — Brighton & Sussex Medical School/Brighton & Sussex Universitys NHS Trust
Locations (1):
- Trevor Mann Baby Unit, Brighton, Sussex, United Kingdom

REFERENCES:
- See also: This is the main clinical trial the study is associated with — http://neocirculation.eu/